CLINICAL TRIAL: NCT00004284
Title: Phase III Randomized, Double-Blind Study of Potassium Phosphate Vs Potassium Citrate for Absorptive Hypercalciuria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Texas (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11703; UTSMC-039510400
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-06

CONDITIONS: Hypercalciuria; Kidney Calculi
Keywords: hypercalciuria; nephrolithiasis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Hypercalciuria; Kidney Calculi; Nephrolithiasis; Rare Diseases; Urogenital Diseases | interventions — Potassium Citrate; potassium phosphate

INTERVENTIONS:
Drug: potassium citrate
Drug: potassium phosphate

SUMMARY:
OBJECTIVES: I. Evaluate the ability of a slow-releasing formulation of neutral potassium phosphate to correct hypercalciuria and prevent recurrent stone formation in patients with absorptive hypercalciuria.

II. Evaluate the safety of this treatment. III. Compare the efficacy of potassium phosphate to that of potassium citrate.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution.

Patients receive potassium phosphate or potassium citrate tablets twice a day for 3 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Absorptive hypercalciuria Intestinal hyperabsorption of calcium, i.e.: Exaggerated calciuric response to oral calcium load OR Fractional calcium-47 absorption greater than 0.61 Calciuria greater than 200 mg/day on random and calcium-restricted diet Normal or high fasting urinary calcium Normal serum calcium Normal serum parathyroid hormone No primary hyperparathyroidism At least 1 calcium oxalate stone within the past 3 years No struvite or carbonate apatite stones No noncalcareous stones No numerous stones making precise quantitation difficult No renal tubular acidosis --Prior/Concurrent Therapy-- No concurrent drug therapy for nephrolithiasis --Patient Characteristics-- Creatinine clearance at least 0.7 mL/min per kilogram No hyperkalemia No hyperphosphatemia No urinary tract infection Other: No predisposition to hyperkalemia, including concurrent use of the following drugs: Potassium-sparing diuretics Angiotensin-converting enzyme inhibitors Nonsteroidal anti-inflammatory drugs No active peptic ulcer disease No chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1995-04

CONTACTS AND LOCATIONS:
Overall Officials: Charles Y. C. Pak, Study Chair — University of Texas